CLINICAL TRIAL: NCT03157375
Title: Rotation of an Intraocular Lens - HOYA Vivinex iSert P261
Acronym: Rot P261
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Menapace, Prof.Dr. Rupert Menapace, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK 1437/2014
Record Dates: First submitted 2017-05-10; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Intraocular Lens
Keywords: IOL, IOL Rotation, Axial Rotation
MeSH Terms: conditions — Intraocular Lymphoma | interventions — Lens Implantation, Intraocular

ARMS (4):
- 0° (Other): Implantation of the intraocular lens Vivinex p261 on axis 0°
  Interventions: Device: Intraocular Lens Implantation
- 45° (Other): Implantation of the intraocular lens Vivinex p261 on axis 45°
  Interventions: Device: Intraocular Lens Implantation
- 90° (Other): Implantation of the intraocular lens Vivinex p261 on axis 90°
  Interventions: Device: Intraocular Lens Implantation
- 135° (Other): Implantation of the intraocular lens Vivinex p261 on axis 135°
  Interventions: Device: Intraocular Lens Implantation

INTERVENTIONS:
Device: Intraocular Lens Implantation

SUMMARY:
Age-related cataract is the main cause of impaired vision in the elderly population worldwide. In the UK, more than half of people who are over 65 years old have some cataract development in one or both eyes. The only treatment that can restore functional visual ability is cataract surgery where the opacified crystalline lens is removed by phacoemulsification and an artificial intraocular lens is implanted. It is estimated that around 10 million cataract operations are performed around the world each year. Cataract operations are generally very successful, with a low risk of serious complications.

During the past two decades, cataract surgery underwent tremendous change and modernisation resulting in today's small incision phacoemulsification surgery and a safe technique with a short rehabilitation time for the patient. Traditional spherical monofocal intraocular lenses (IOLs) restore best-corrected vision and may lessen the need for spectacles. These IOLs correct only the spherical portion of the total refractive error and do not correct corneal astigmatism. Astigmatism is a visually disabling refractive error affecting the general population, especially those with cataract. At least 15% to 20% of cataract patients have 1.5 diopters (D) or more of corneal or refractive astigmatism. With increased patient expectations, the trend is not only to remove the cataract but also to address the problem of pre-existing astigmatism at the time of surgery.

Surgical-induced astigmatism can be reduced by smaller incisions, i.e. microincision cataract surgery (MICS), which by definition is surgery performed through incisions smaller than 2.0 mm, reducing the need for suturing. This results in better corneal optical quality, thus improving visual outcomes. There are also other surgical options to correct preexisting astigmatism during cataract surgery like: selectively positioning of the phacoemulsification incision; astigmatic keratotomy with corneal or limbal relaxing incisions; excimer laser refractive procedures such as photorefractive keratectomy, laser in situ keratomileusis, and laser-assisted subepithelial keratectomy; or implanting pseudophakic toric posterior chamber intraocular lenses (IOLs).

Toric IOLs have been shown to result in good visual and refractive outcomes. Combined with MICS, these IOLs can allow effective correction of cylindrical errors intraoperatively, improving visual quality and thus leading to spectacle independence. Plate haptic and loop haptic toric IOLs have been considered for about a decade but have been associated with postoperative rotational instability. Rotation of a toric lens from its intended orientation degrades its corrective power, with approximately 3.3% loss of cylindrical power for every degree off axis. A misorientation of approximately 30° negates the effectiveness of astigmatic correction, and a misorientation of more than 30° may induce additional astigmatism. Although some patients are asymptomatic despite induced astigmatism, others experience symptoms such as blurred or distorted vision, headache, fatigue, eyestrain, squinting, or eye discomfort. Thus, IOL orientation stability is an essential goal in toric IOL design.

RATIONALE

The purpose of this study is to assess the axial IOL rotation and optical quality (refraction, visual acuity, contrast sensitivity, decentration and tilt) and capsular bag reaction after micro-incision surgery with an IOL implantation in cataract patients - HOYA Vivinex iSert® model P261.

ELIGIBILITY:
Inclusion Criteria:

* Uni- or bilateral age-related cataract necessitating phacoemulsification extraction and posterior IOL implantation
* Need for spherical IOL correction between 15.00 and 25.00 D
* Pupil dilation of ≥ 6.5 mm
* Age 50 and older

Exclusion Criteria:

* Corneal abnormality
* Pseudoexfoliation
* Preceding ocular surgery or trauma
* Uncontrolled glaucoma
* Proliferative diabetic retinopathy
* Iris neovascularization
* History of uveitis/iritis
* Microphthalmus
* Recurrent intraocular inflammation of unknown etiology
* Blind fellow eye
* Uncontrolled systemic or ocular disease
* Pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-10-06; Primary Completion 2015-10-02 (Actual); Study Completion 2015-10-02 (Actual)

PRIMARY OUTCOMES:
Change of axial intraocular lens position | 7 months
  Change in axial intraocular lens position from end of surgery (baseline axis) to 4-7 months (end of study visit)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, Vienna, Austria